CLINICAL TRIAL: NCT03535168
Title: Two-part, Double-blind, Placebo-controlled, Randomized, Parallel-group Study: (Part 1) in Healthy Male Subjects to Assess Safety and Tolerability of Ascending Repeated Oral Doses of BAY1902607 Including Its Effect on the Pharmacokinetics of a Sub-therapeutic Dose of Midazolam (MDZ), Followed by (Part 2) a Two-way Crossover Administration of Four Different Doses of BAY1902607 in Patients With Refractory Chronic Cough to Assess Safety, Tolerability and Efficacy for Proof of Concept
Brief Title: Repeat Doses of BAY1902607 in Healthy Males and Proof of Concept in Chronic Cough Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19430; 2018-000129-29 (EudraCT Number)
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Cough
Keywords: Healthy volunteers
MeSH Terms: conditions — Cough | interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: Part 1: Sequential parallel-group Part 2: Two-arm crossover
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Dose 1 of BAY1902607 (Experimental): Part 1: From Day 1 until Day 12 the dose 1 of BAY1902607 will be given twice daily in approximately 12 hour intervals. On Day 0 and Day 13, dose 1 of BAY1902607 will be given only once.
  Interventions: Drug: BAY1902607; Drug: Midazolam
- Dose 2 of BAY1902607 (Experimental): Part 1: From Day 1 until Day 12 the dose 2 of BAY1902607 will be given twice daily in approximately 12 hour intervals. On Day 0 and Day 13, dose 2 of BAY1902607 will be given only once.
  Interventions: Drug: BAY1902607; Drug: Midazolam
- Dose 3 of BAY1902607 (Experimental): Part 1: From Day 1 until Day 12 the dose 3 of BAY1902607 will be given twice daily in approximately 12 hour intervals. On Day 0 and Day 13, dose 3 of BAY1902607 will be given only once.
  Interventions: Drug: BAY1902607; Drug: Midazolam
- Matching placebo (Experimental): Part 1: From Day 1 until Day 12 the matching placebo will be given twice daily in approximately 12 hour intervals. On Day 0 and Day 13, matching placebo will be given only once.
  Interventions: Drug: Matching placebo; Drug: Midazolam
- BAY1902607+Matching Placebo (Experimental): Part 2:
  Randomized crossover design in cough patients 4 different doses of BAY1902607+matching placebo
  Interventions: Drug: BAY1902607; Drug: Matching placebo
- Matching Placebo+BAY1902607 (Experimental): Part 2:
  Randomized crossover design in cough patients Matching placebo+4 different doses of BAY1902607
  Interventions: Drug: BAY1902607; Drug: Matching placebo

INTERVENTIONS:
Drug: BAY1902607 — 3 different doses over the course of part 1 and 4 different doses over the course of part 2.
  Arms: BAY1902607+Matching Placebo; Dose 1 of BAY1902607; Dose 2 of BAY1902607; Dose 3 of BAY1902607; Matching Placebo+BAY1902607
Drug: Matching placebo — Matching placebo for BAY1902607
  Arms: BAY1902607+Matching Placebo; Matching Placebo+BAY1902607; Matching placebo
Drug: Midazolam — Part 1: The subjects will initially (Day -1) receive a sub-therapeutic dose of 1 mg midazolam as solution in the morning.
  Arms: Dose 1 of BAY1902607; Dose 2 of BAY1902607; Dose 3 of BAY1902607; Matching placebo

SUMMARY:
The primary objectives of this study:

* To investigate the safety and tolerability of ascending repeated oral doses of BAY1902607 in healthy subjects (Part 1).
* To investigate the effect of BAY1902607 on the pharmacokinetics (PK) of a sub-therapeutic 1 mg dose of midazolam (Part 1).
* To investigate the safety, tolerability and efficacy of BAY1902607 in patients with refractory chronic cough (Part 2).

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* Male; healthy according to complete medical history, including the physical examination, vital signs (blood pressure, heart rate), 12-lead ECG, clinical laboratory tests
* Age: 18-45 years (inclusive) at the first screening visit
* Non-smoker for at least 6 months and with a pack year history of equal to or less than 5 years
* Subjects, who are sexually active and have not been surgically sterilized, must agree to use two reliable and acceptable methods of contraception simultaneously, when having sexual intercourse with women of childbearing potential (one method used by the subject, one method used by the partner) during the study and for 90 days after receiving the investigational medicinal product, and not to act as sperm donor for 90 days after dosing. [Acceptable methods of contraception include for example: (a) condoms (male or female) with or without a spermicidal agent, (b) diaphragm or cervical cap with spermicide, (c) intrauterine device, (d) hormone-based contraception]

Part 2:

* Age: ≥18 years at the first screening visit
* Refractory chronic cough for at least one year that has been shown to be unresponsive to treatment of cough according to the 2006 British Thoracic Society (BTS) guideline
* Score of ≥ 40 mm on the Cough Severity visual analogue scale (VAS) at screening
* For female patients:

Confirmed post-menopausal woman (defined as exhibiting spontaneous amenorrhea for at least 12 months before screening or as exhibiting spontaneous amenorrhea for 6 months before screening with documented serum follicle-stimulating hormone (FSH) levels > 40 mIU/mL) or Woman without childbearing potential based on surgical treatment at least 6 weeks before screening, such as bilateral tubal ligation, bilateral oophorectomy with or without hysterectomy (documented by medical report verification) or Woman of childbearing potential that agrees to use two reliable and acceptable methods of contraception simultaneously (one method used by the study patient and one method used by the partner) during the study and for at least 31 days (1 average menstrual cycle of 28 days plus approx. 5 half-lives of BAY 1902607) after the last dose. In addition during the study and for at least 31 days after the last dose women of child bearing potential are not allowed to donate oocytes.

Exclusion Criteria:

Part 1:

* Relevant diseases potentially interfering with the study objectives (e.g. respiratory diseases) within the four weeks before screening or between screening and randomization
* Any febrile illness within the four weeks before screening or between screening and randomization
* Medical history of hypogeusia/dysgeusia or the subject has a dysfunction in his ability to taste, as revealed by the taste-disturbance questionnaire during screening and the predose procedures

Part 2:

* FEV1(Forced Expiratory Volume in 1 second) or FVC(Forced Vital Capacity ) of less than 60% of predicted normal, at screening
* History of upper or lower respiratory tract infection or recent significant change in pulmonary status within the 4 weeks before screening
* Current smoking habit or history of smoking within the 6 months before the screening visit
* History of smoking (at any time) for more than 20 pack-years in total (20 cigarettes per pack)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Treatment-Emergent Adverse Events (TEAEs) by Severity in Part 1 | Approximately 5 weeks
Number of subjects with Treatment-Emergent Adverse Events (TEAEs) by Severity in Part 2 | Approximately 12 weeks
AUC of midazolam without BAY1902607 | At Day -1
  Part 1
AUC of midazolam in combination with BAY1902607 | At Day 13
  Part 1
Cmax of midazolam in combination with BAY1902607 | At Day 13
  Part 1
Cmax of midazolam without BAY1902607 | At Day -1
  Part 1
Number of Coughs Experienced by the Patient Within a 24-hour Period (24- hour cough count/hour) in Part 2 | 24 hours
  Part 2: Coughs monitored by VitaloJAK cough recorder (Vitalograph)

CONTACTS AND LOCATIONS:
Locations (8):
- Netherlands (2):
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - Isala, Zwolle
- United Kingdom (6):
  - Queen's University, Belfast, Antrim
  - Birmingham Heartlands Hospital, Birmingham, West Midlands
  - Castle Hill Hospital, Cottingham
  - King's College Hospital - NHS Foundation Trust, London
  - Medicines Evaluation Unit, Manchester
  - University Hospital of South Manchester, Manchester

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Friedrich C, Francke K, Birring SS, van den Berg JWK, Marsden PA, McGarvey L, Turner AM, Wielders P, Gashaw I, Klein S, Morice AH. The P2X3 receptor antagonist filapixant in patients with refractory chronic cough: a randomized controlled trial. Respir Res. 2023 Apr 11;24(1):109. doi: 10.1186/s12931-023-02384-8. PMID 37041539
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/